CLINICAL TRIAL: NCT00539357
Title: A Pilot Study of Cranial Electrotherapy Stimulation[CES] for Generalized Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-08-121-02
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Generalized Anxiety Disorder
Keywords: Cranial Electrostimulation Therapy
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All patients self-administered stimulation for 60 consecutive minutes each day. Participants self-administered the treatment for a period of 6 weeks, 7 days a week between the hours of 15:00 and 19:00. Assessments took place every 2 weeks during the treatment period.
  Interventions: Device: Cranial electrotherapy stimulation (CES)

INTERVENTIONS:
Device: Cranial electrotherapy stimulation (CES) — Cranial electrotherapy stimulation (CES) is a noninvasive procedure that involves applying a pulsed, low-amplitude electrical current to the head using electrodes placed on the earlobes. Cranial electrotherapy stimulation CES received U.S. Food and Drug Administration (FDA) approval for the treatment of insomnia, depression, and anxiety in 1979.
  Other Names: Alpha-Stim Stress Control System (SCS)

SUMMARY:
Cranial electrotherapy stimulation(CES) is a noninvasive procedure that has been used for decades in the United States to treat anxiety, depression, and insomnia in the general population. Whether CES is an effective treatment for patients with a DSM-IV diagnosis of generalized anxiety disorder (GAD) has not previously been explored. The goal of this study was is to evaluate the efficacy of CES in alleviating anxiety in patients with DSMIV-diagnosed GAD. Specifically our hypothesis was that CES would demonstrate possible efficacy in reducing symptoms associated with GAD from baseline to end of trial, as determined by: (1) change from baseline in the Hamilton Anxiety Scale (HAM-A) total score. a.) the proportion of responders (much or very much improved) as assessed by the CGI Improvement ratings by visit b.) the proportion of responders (50% reduction from total HAM A baseline score) according to the HAM A scores by visit c.) the proportion of patients in remission (HAM A score ≤7) by visit

DETAILED DESCRIPTION:
This study utilized a 6-week open-label design to test CES in the treatment of GAD. The study was funded by Saban Family foundation. The devises were provided by Electromedical Products Inc. (EPI) which is a technology company manufacturing the cranial stimulators. This company has no relationship with any of the investigators of the study. There are no explicit or implicit conflicts of interest. Participants were recruited from August 2005 to March 2006 from the UCLA Anxiety Disorders Program at the Semel Institute for Human Behavior. Permission from UCLA's Institutional Review Board was obtained to conduct this study. All eligible subjects provided approved written consent prior to the initiation of any study related procedure.

Patient Selection: Male or female outpatients aged 18 to 64 years were eligible if they had a current diagnosis of GAD. At screening, GAD diagnosis was confirmed by conducting the MINI interview.(Sheehan, Lecrubier et al. 1998) Patients had to have a score ≥ 16 on the Hamilton Anxiety Rating Scale (HARS) and < 17 on the 17-Item Hamilton Depression Rating Scale (HDRS) at baseline to be considered for enrollment.(Hamilton 1959; Hamilton 1960) Lower then usual HARS were permitted to include milder cases of GAD. Patients were excluded if they had a primary diagnosis meeting DSM-IV criteria for any other Axis I disorder other than GAD, as were patients who met DSM-IV criteria for mental retardation, any pervasive developmental disorder or neurological impairment. Also excluded were those with a recent (6 months) history or current diagnosis of drug or alcohol dependence or abuse, current suicidal ideation and/or history of suicide attempt or any personality disorder of sufficient severity to interfere with participation in the study. Other exclusion criteria included a history or presence of a medical disease that might compromise the study or be detrimental to the patient. Women who were pregnant or breastfeeding and women of childbearing potential who were not practicing a reliable form of contraception were also excluded from the study and the use of any psychotropic medication. Patients were permitted to be on a stable, therapeutic dose of SSRI or SNRI if they were taking their medications for at least 3 month and were still symptomatic after at least 3 months of treatment. Patients who used PRN as-needed benzodiazepines were permitted to enter the study if their use of the medications did not exceed two times per week. Women who were pregnant or breastfeeding and women of childbearing potential who were not practicing a reliable form of contraception were also excluded from the study. Study visits were conducted at baseline and at the end of 3 and 6 weeks of treatment. Patients who met all of the eligibility criteria at baseline were enrolled and administered CES treatment.

Results: Fifteen subjects expressed interest in the study and engaged in an initial telephone screen. Eight percent (n=3) of participants were deemed ineligible to participate. Reasons for ineligibility included age (n=1; 3%) and psychiatric co morbidity (n=2; 6%). Twelve subjects enrolled and received CES treatment. The mean age of the sample was 42.83±10.7 years. Of the twelve individuals enrolled in the study 9 (75%) were female and 3 (25%) were male. Five participants (41.6%) had been taking psychotropic medications for at least 3 months prior to enrollment and continued throughout the study; two participants took venlaflaxine and the remaining 3 patients took benzodiazepines on an as-needed basis no more than twice a week (2 took alprazolam, and 1 took lorazepam). Overall, 75% of patients (n=9) completed the study. Three subjects discontinued after baseline due to adverse events, including dizziness (n=2) and headache (n=1). A significant change (11.5 points) was found from baseline to endpoint in HARS scores (t= 8.59 p= 0.001). The mean change from baseline was significant after 2 weeks of treatment and continued to increase over time. At endpoint, 6 (66%) of 9 patients had a 50% decrease on HARS and a score of 1 or 2 on CGI improvement, and were considered responders to treatment. An additional patient improved but did not meet criteria for response. Mean HDRS score changed from 10.5±15.01 at baseline to 6±3.64 at endpoint (t= 3.01, p=0.01). A significant change was also found from baseline (30.3±11.49) to endpoint (23.3±6.76) in UCLA 4D Anxiety Subscale scores (t=2.63, p= 0.03).

Results of the current study demonstrate a significant improvement with CES, with a decrease in HARS score similar to that found in clinical trials with antidepressant and anxiolytic medications .(Katz, Reynolds et al. 2002; Rickels and Rynn 2002; Pollack, Meoni et al. 2003; Sheehan and Mao 2003; Bielski, Bose et al. 2005; Brawman-Mintzer, Knapp et al. 2006; Dhillon, Scott et al. 2006). The effect size is 2.4 appears to be very large. However, it is expected in an open trial where some part of the parts of the effect could be due to placebo response. The above cited studies had an effect size for placebo ranging from 0.74 to approximately 1.72. Most of the recent pharmacological studies in GAD observed a large placebo response which makes it imperative to conduct placebo-controlled or sham-controlled study to fully evaluate the treatment effect in this population (Rickels and Rynn 2002)

The patients generally liked the treatment and 3 of them continued to use the devise after the experiment was over and purchased their own CES stimulator. However, 3 of the subject experience the side effects which caused them to withdraw prematurely from the study. Presence of side effects in some of the patients could be the sign of some physiological effect in these patients which needs to be studied in future studies.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female outpatients age 18 to 65 years, inclusive
2. The subject meets DSM-IV criteria for Generalized Anxiety Disorder as determined by the MINI
3. Sexually active female patients of childbearing potential must be practicing at least one or more the following methods of contraception during the study: intrauterine device (IUD), barrier method in combination with a spermicide, oral/hormonal contraception or abstinence. Female patients of childbearing potential must have a negative pregnancy test prior to receiving study drug.
4. Written informed consent must be obtained from the subject prior to study participation.
5. The subject is in good medical health or with chronic medical conditions which are currently stable.
6. No current abuse of alcohol or other substance.
7. The subject has a total score of 20 or more on the Hamilton Anxiety Scale (HAMA) at screening.
8. The subject has a Clinical Global Impression (CGI) Severity score of 4 or more at screening.

Exclusion Criteria:

1. The subject meets DSM-IV criteria for an Axis I diagnosis (other than GAD) as the primary diagnosis (i.e., schizophrenia, mood disorder, psychosis, anorexia nervosa) as determined by the MINI.
2. The subject is clinically judged by the investigator to be at risk for suicide or is acutely suicidal as objectively measured by the MINI and MSE.
3. The subject is clinically judged by the investigator to be at risk for homicide or is acutely homicidal as objectively measured by the MINI and MSE.
4. The subject has a psychiatric condition that would require inpatient, or partial psychiatric hospitalization.
5. Seizure disorders.
6. Significant history of medical disease (i.e. cardiovascular, hepatic (e.g. cirrhosis, hepatitis B or C) renal, gynecological, musculoskeletal, neurological, gastrointestinal, metabolic, hematological, endocrine, cancer with a metastatic potential or progressive neurological disorders) which could impair reliable participation in the trial or necessitate the use of medication not allowed by this protocol.
7. The subject is pregnant, planning to become pregnant, or nursing. If a subject becomes pregnant, she will be discontinued immediately and followed appropriately.
8. Concomitant therapy with another investigational drug, or participation in an investigational drug study within one month prior to entering this study.
9. Current psychotherapeutic treatment except for treatment with Specific Reuptake Inhibitor (SSRIs) medications which include: Fluoxetine (Prozac), Paroxetine (Paxil), Sertraline (Zoloft), Luvox (Fluvoxamine), and Citalopram. Potential subjects may remain on one of the SSRI medications provided that he or she has been on a stable dose for at least 4 weeks prior to entering this study; this dose remains stable throughout the remainder of this study; and it can be determined that this medication is not exacerbating the anxiety symptoms.
10. History of poor compliance or in the Investigator's judgment patients any subject whose treatment as an outpatient would be clinically contraindicated
11. The subject has attempted suicide one or more times within the past twelve months
12. The subject has a Hamilton Depression Rating Scale (HAM-D) score above 38 which suggests a moderate to severe clinical level of depressive symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-08; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The Hamilton Anxiety Rating Scale (HAM-A) | at baseline and after 3 and 6 weeks of treatment

SECONDARY OUTCOMES:
the Clinical Global Impression Improvement CGI-I scale (beginning at week 2), the 17-item Hamilton Rating Scale for Depression, Patients Global Impressions-Improvement ande the Four-Dimensional Anxiety and Depression Scale | baseline, and after 3 and 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bystritsky, MD, Principal Investigator — University of California, Los Angeles

REFERENCES:
- [Derived] Bystritsky A, Kerwin LE, Feusner JD. A preliminary study of fMRI-guided rTMS in the treatment of generalized anxiety disorder: 6-month follow-up. J Clin Psychiatry. 2009 Mar;70(3):431-2. doi: 10.4088/JCP.08l04641. No abstract available. PMID 19317960
- [Derived] Bystritsky A, Kaplan JT, Feusner JD, Kerwin LE, Wadekar M, Burock M, Wu AD, Iacoboni M. A preliminary study of fMRI-guided rTMS in the treatment of generalized anxiety disorder. J Clin Psychiatry. 2008 Jul;69(7):1092-8. doi: 10.4088/jcp.v69n0708. PMID 18572984
- [Derived] Bystritsky A, Kerwin L, Feusner J. A pilot study of cranial electrotherapy stimulation for generalized anxiety disorder. J Clin Psychiatry. 2008 Mar;69(3):412-7. doi: 10.4088/jcp.v69n0311. PMID 18348596